CLINICAL TRIAL: NCT03521739
Title: A National Registry for the Association of Synchronous Four-limb Blood Pressure and Pulse Wave Velocity With Cardiovascular Events in China
Brief Title: Association of Synchronous Four-limb blOod pRessure and Pulse Wave velocIty With Cardiovascular Events
Acronym: ASORPWICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Xiongjing Jiang, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2018-993
Record Dates: First submitted 2018-04-11; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Blood Pressure; Pulse Wave Analysis; Ankle Brachial Index; Patient Outcome Assessment
Keywords: blood pressure; pulse wave velocity; ankle brachial index; cardiovascular events

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A multicenter prospective registry planned to recruit more than 100 000 patients 50 years old and older was carried out in China. This primary purpose of this study was to evaluate the association of synchronous four-limb blood pressure and pulse wave velocity with cardiovascular events. The secondary purpose was to evaluate the incidence rate,prevalence rate, value of diagnosis for peripheral arterial occlusive disease, and to follow up the effects of revascularization on cardiovascular events.

DETAILED DESCRIPTION:
Although many studies with the correlation between synchronous four-limb blood pressure and pulse velocity measurement and cardiovascular outcomes have existed currently, the sample sizes are relatively small and the data on Chinese populations are lacking.Therefore, a multicenter prospective registry planned to recruit more than 100 000 patients aged 50 years old and older was carried out in China. This primary purpose of this study was to evaluate the association of synchronous four-limb blood pressure and pulse wave velocity with cardiovascular events in chinese populations. The secondary purpose was to evaluate the incidence rate,prevalence rate, value of diagnosis for peripheral arterial occlusive disease, and to follow up the effects of revascularization on cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years old at the time of informed consent
2. Chinese populations in hospital, community and physical examination center

Exclusion Criteria:

1. Patients with lack of limb,malformation of limbs, severe limb trauma or infection.
2. Serious organic disease affecting the quality of life, such as tumors, massive cerebral infarction, uremia, and etc.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese populations with age ≥ 50 years old at the time of informed consent in hospital, community and physical examination center
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiovascular events (cardiovascular death,myocardial infarction, heart failure, stroke, renal failure, aortic dissection) | From date of enrollment until the date of first documented cardiovascular events or date of death from any cause, whichever came first, assessed up to 12 months

SECONDARY OUTCOMES:
Incidence of cardiovascular events (cardiovascular death,myocardial infarction, heart failure, stroke, renal failure, aortic dissection) | Measured at 6 months, 24 months and every 12 months thereafter from date of enrollment until the date of first documented cardiovascular events or date of death from any cause, whichever came first, assessed up to 60 months
Incidence of death from any cause | Measured at 6 months, 12 months and every 12 months thereafter from date of enrollment until the date of first documented death from any cause, assessed up to 60 months
Incidence of peripheral arterial disease | Measured at 6 months, 12 months and every 12 months thereafter from date of enrollment until the date of first documented four-limb peripheral arterial disease or date of death from any cause, whichever came first, assessed up to 60 months
Incidence of limb gangrene | Measured at 6 months, 12 months and every 12 months thereafter from date of enrollment until the date of first documented gangrene caused by peripheral arterial disease or date of death from any cause,whichever came first, assessed up to 60 months
Incidence of amputation | Measured at 6 months, 12 months and every 12 months thereafter from date of enrollment until the date of first documented amputation caused by peripheral arterial disease or date of death from any cause, whichever came first, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiongjing Jiang, MD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (19):
- China (19):
  - Beijing Renhe Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Daping Hospital, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The Eighth Affiliated Hospital of Sun Yat-sen University, Shenzhen, Guangdong
  - Kailuan General Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The General Hospital of Shenyang Military, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Xi'an NO.3 Hospital, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Zhejiang Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] An X, Dong H, Deng Y, Chen Y, Zou Y, Zhang W, Jiang X. Evaluation of the role of combining inter-arm systolic pressure difference and derivatives of pulse volume recording in detecting subclavian artery stenosis. Front Cardiovasc Med. 2022 Sep 15;9:962610. doi: 10.3389/fcvm.2022.962610. eCollection 2022. PMID 36186962